CLINICAL TRIAL: NCT04042870
Title: Effect of Sukshma Vyayama Joint Loosening Yoga on Aromatase Inhibitor-Induced Arthralgia in Post-Menopausal Breast Cancer Survivors: A Feasibility Study Conducted on Facebook
Brief Title: Effect of Sukshma Vyayama Yoga on Aromatase Inhibitor-Induced Arthralgia in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AshtaYoga, LLC (Industry)
Collaborators: Columbia University (Other); Swami Vivekananda Yoga Anusandhana Samsthana (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AI Yoga Study on Facebook - 1
Record Dates: First submitted 2019-07-14; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Yoga; Aromatase Inhibitor; Arthralgia; Sukshma Vyayama
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Intervention Model Description: Pre / Post Single Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Joint Loosening Yoga (Experimental): Yoga Intervention. Dose: 15 minutes, M-F for 4-weeks.
  Interventions: Behavioral: Joint Loosening Yoga

INTERVENTIONS:
Behavioral: Joint Loosening Yoga — Sukshma Vyayama Joint Loosening Yoga was practiced Monday - Friday for four weeks. Each session included twelve joint loosening exercises performed in a chair, each performed 10 times with mindful awareness of physical movements and breath synchronization. Sessions lasted 15 minutes.

SUMMARY:
The purpose of this study is to investigate the efficacy of sukshma vyayama joint loosening yoga in improving aromatase inhibitor-induced arthralgia in post-menopausal breast cancer survivors and secondarily, to evaluate the feasibility of delivering the intervention on Facebook.

DETAILED DESCRIPTION:
Cancer survival rates are improving in the United States but this increased survivorship is offset by persistent treatment related symptoms, particularly for post-menopausal breast cancer survivors treated with aromatase inhibitor (AI) hormonal therapy. AI therapy is well known to cause arthralgia that can compromise a woman's quality of life. National Comprehensive Cancer Center Network (NCCCN) guidelines for breast cancer treatment recommend that post-menopausal women with estrogen receptor-positive tumors receive aromatase inhibitors, e.g., anastrozole (Arimidex), letrozole (Femara) or exemestane (Aromasin) as a key part of treatment to lower the risk of breast cancer recurrence, breast cancer in the opposite breast, and death from breast cancer. Estrogen receptor-positive breast cancer represents almost 50% of all newly diagnosed cases of breast cancer. Currently, AIs are prescribed for five to ten years. The length of this treatment, coupled with difficult arthritic side effects can make it difficult for patients to complete therapy. Arthralgia occurs in up to 50% of breast cancer survivors treated with AIs and is the most common reason for poor AI adherence. Up to 50% of patients do not take AIs as prescribed and up to 20% will become non-compliant with treatment within the first year due to pain and discomfort. To get the most benefit out of hormone therapy, however, patients must take the full course of treatment. Both non-adherence and early discontinuation of AIs have been shown to be independent predictors of mortality. Women who complete the full course have better survival than those who do not. Given the efficacy of AIs in preventing breast cancer recurrence, and the proportion of women who discontinue these drugs because of adverse events, interventions to improve adverse effects are important.

This study investigated the efficacy of sukshma vyayama joint loosening yoga in reducing and improving aromatase inhibitor-induced joint pain and achiness in post-menopausal breast cancer patients, and evaluated the feasibility of delivering the intervention on Facebook. Hypothesis: Given global disparities in healthcare, being able to safely deliver evidence-based yoga interventions via the internet is important.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal breast cancer survivors undergoing treatment with aromatase inhibitor hormonal therapy with self-reported arthralgia
* Must have initiated anastrazole, exemestane, or letrozole within 30 days of baseline assessment
* 35-70 years old
* Must be available during the dates of the study and willing to participate in the study
* Must have access to computer, tablet or smart phone and Internet connection
* Must be a member of Facebook
* Eligible if their arthralgia started after initiation of an AI or if they had preexisting joint pain that was exacerbated by AI use
* English speaking

Exclusion Criteria:

* Non English-speaking
* Physically unable to perform the intervention

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with estrogen receptor-positive breast cancer prescribed and currently taking aromatase inhibitor therapy.
Enrollment: 38 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Arthralgia Inventory (PRAI) Measure for Joint Arthralgia | Baseline and Four weeks
  The Patient-Reported Arthralgia Inventory measures self-reported pain intensity in 16 specific joints over the past 7 days. This questionnaire consists of 16 questions answered on a 0 to 10 scale (0 = no pain at all; 10 = worst pain you can imagine) with a min of 0 and a max of 160. Higher scores indicate more pain.
Change in Brief Pain Inventory Short Form (BPI SF) Measure for Body Pain | Baseline and Four weeks
  The Brief Pain Inventory Short Form measures self-reported pain intensity in the body in the last 24-hours. This questionnaire consists of 8 questions (4 on pain quality) answered on a scale 0-10 (0 = no pain; 10 = pain as bad as you can imagine) with a min of 0 and a max of 40. Higher scores indicate more pain.
Change in Brief Pain Inventory Short Form (BPI SF) Measure for Quality of Life | Baseline and Four weeks
  The Brief Pain Inventory Short Form measures self-reported QoL in the last 24-hours. This questionnaire consists of 7 questions answered on a scale 0-10 (0 = does not interfere; 10 = completely interferes) with a min of 0 and a max of 70. Higher scores indicate lower QoL.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Measure for Pain, Stiffness, and Physical Function of Knee and Hip | Baseline and Four weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index measures self-reported pain, stiffness, and functional limitation of knee and hip during activity in the last 48-hours. This questionnaire consists of 24 questions answered on a scale 0-4 (0 = none; 4 = extreme). Measures include five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores indicate greater pain, stiffness, and functional limitation.
Change in Disability of the Arm, Shoulder and Hand (DASH) Measure of Ability to Use Arm, Shoulder, and Hand | Baseline and Four weeks
  The Disability of the Arm, Shoulder and Hand tool measures self-reported ability to do daily activities in the last week and impact on QoL. The questionnaire consists of 30 questions answered on a scale 1-5 (1 = no difficulty; 5 = unable) with a min of 30 and a max of 150. Measures include 21 items for daily functional activity (score range 30-105), two for interference with social or work activity (score range 2-10), five for pain and discomfort (score range 5-25), one for sleep (score range 1-5), and one for confidence (score range 1-5). Higher scores indicate greater pain and disability.

SECONDARY OUTCOMES:
Effectiveness of Delivering Intervention on Facebook | Four Weeks
  Measure whether sufficient numbers of subjects enroll in order to complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Leibel, MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leibel L, Metri K, Prasad R, Mears JG, Effect of Sukshma Vyayama on Aromatase Inhibitor-Induced Arthralgia in Post-Menopausal Breast Cancer Survivors: A Feasibility Study Conducted on Facebook, J Clin Oncol 37, 2019 (suppl; abstr e23129)